CLINICAL TRIAL: NCT04522804
Title: A Pilot Study of Psilocybin Enhanced Group Psychotherapy in Patients With Cancer
Brief Title: Study of Psilocybin Enhanced Group Psychotherapy in Patients With Cancer
Acronym: HOPE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI131965
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental): Subjects will participate in a total of seven group sessions. There will be 4 or 6 subjects per group and one therapist will be assigned to each subject for a total of 4 or 6 therapists. In addition, there will be one Group Leader that will facilitate the group sessions. Group sessions will occur once per week for approximately five weeks. The first three sessions are "Preparatory" sessions followed by three "Integration" sessions. During the week following the third Preparatory session and prior to the first Integration session, participants will participate in a psilocybin session.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is a classic psychedelic of medium duration that is well-tolerated and has a documented safety and efficacy record that makes it uniquely well-suited to the existential issues that arise in this patient population. Psilocybin has been described as an 'existential medicine' given patient testimonials as to its acute and lasting effects on interpersonal connection, ability to more deeply engage with meaningful activities and relationships, dramatic reductions in fear of death, and a renewed sense of well-being.

SUMMARY:
This pilot project is an open-label trial that will offer psilocybin in a group format to assess the feasibility of offering psilocybin therapy in a group setting with a decreased therapist to subject ratio. Study intervention will involve a group of six patients with one therapist per subject for a 1:1 ratio, thus significantly reducing the total number of therapist hours per subject compared to standard individual therapy protocols.

Two groups of six will be treated on this trial. After the enrollment and treatment of the first group of six patients, accrual will be placed on hold to ensure subject safety. If stopping rules are not met (Section 11), the next group of six patients will be enrolled and treated on study.

The study intervention will include a total of seven group therapy sessions including three 2-hour preparatory sessions, one 8-hour psilocybin session, and one two-hour integration session. The group therapy sessions will occur on a weekly basis, followed one week later by the psilocybin session. The first integration group session will occur 1-2 days following the psilocybin session.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 25 years old.
* Current diagnosis of cancer and undergoing treatment for their cancer or completed treatment within ≤ 26 weeks of study registration.
* Life expectancy ≥ 3 months.
* Current DSM-V diagnosis of a depression disorder including adjustment disorder with disturbance of mood.
* Not taking regularly scheduled medications to treat depression and/or anxiety, including benzodiazepines, for at least 4 weeks prior to initiation of the study.
* Fluent in English.
* Have a high school or equivalent (e.g., GED) level of education. Volunteers without a high school or equivalent education must demonstrate reading literacy and comprehension sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* ECOG Performance Status ≤ 2.
* Have a support person that would be able to escort the subject home on the evening of the psilocybin dosing session.
* Adequate liver function as defined as:

  * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) unless elevated bilirubin is related to Gilbert's Syndrome.
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
* For female subjects: Negative pregnancy test and agreement to use highly effective contraception (as described in Section 7.2) or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, ondansetron, cannabis, and non-routine PRN medications within 24 hours of each psilocybin administration. Exceptions include daily use of caffeine, nicotine, and opioid pain medication (see Section 6.2.2).
* Agree that for one week preceding the psilocybin session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Agree not to use nicotine for at least 2 hours before the psilocybin administration.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of the psilocybin session. If the subject does not routinely consume caffeinated beverages, he or she must agree not to do so on the day of psilocybin administration.
* Subjects requiring opioid use for pain are on a stable pain management regimen. Long-acting opioid medications (e.g., oxycodone sustained-release, morphine sustained release) will be allowed if the last dose occurred at least 6 hours before psilocybin administration; such medication will not be taken again until at least 6 hours after psilocybin administration.

Exclusion Criteria:

* Positive screening SARS-CoV2 (COVID-19) test, symptoms of COVID-19, or contact with someone who has tested positive for COVID-19.
* Prior systemic antidepressants, anti-psychotic, or anxiolytic medication within four weeks prior to study initiation.
* Personal history or immediate family members with schizophrenia, bipolar affective disorder, delusional disorder, schizoaffective disorder, psychosis, or other psychotic spectrum illness.
* Currently meeting DSM-V criteria for Dissociative Disorder, or other psychiatric conditions judged to be incompatible with the establishment of rapport or safe exposure to psilocybin.
* Currently meeting DSM-V criteria for Cluster B Personality Disorder.
* Current or history within the last two years of meeting DSM-V criteria of substance use disorder (excluding caffeine and nicotine).
* Severe depression requiring immediate standard-of-care treatment e,g.,hospitalization.
* Suicidal ideation with active intent or plan to act on suicidal thoughts as assessed by the treating investigator.
* Cancer with known CNS involvement, or other major CNS disease.
* Involvement in another investigational product for the treatment of cancer.
* Known paraneoplastic syndrome or other ectopic hormone production by a tumor.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class III or IV
    * Unstable angina pectoris, cardiac hypertrophy, cardiac ischemia, myocardial infarction
    * Uncontrolled hypertension at time of enrollment (BP>140 systolic or 90 diastolic), coronary artery disease, artificial heart valve
    * Prolonged or congenital long QT syndrome (≥480 ms), serious cardiac arrhythmias, tachycardia, a clinically significant screening ECG abnormality
  * Renal insufficiency as defined as creatinine clearance < 40 mL/min calculated by Cockcroft-Gault formula:

    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
    * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
  * Hepatic disorders:

    * Active infection including hepatitis B (known positive HBV surface antigen (HBsAg) result) or hepatitis C.
    * Note: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [patients may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Known prior severe hypersensitivity to investigational product or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.3.2. A washout period of prohibited medications for a period of at least five half-lives should occur prior to study registration.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by severity | 8 months
  assess the safety of psilocybin in patients with a cancer diagnosis or hematologic malignancy.
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by duration | 8 months
  assess the safety of psilocybin in patients with a cancer diagnosis or hematologic malignancy.
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by relationship to study treatment. | 8 months
  assess the safety of psilocybin in patients with a cancer diagnosis or hematologic malignancy.
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by seriousness | 8 months
  assess the safety of psilocybin in patients with a cancer diagnosis or hematologic malignancy.
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by type | 8 months
  assess the safety of psilocybin in patients with a cancer diagnosis or hematologic malignancy.
recruitment of patients with cancer diagnosis or hematologic malignancy | 18 months
  assess the feasibility to recruit patients with a cancer diagnosis or hematologic malignancy
Enrollment of patients with a cancer diagnosis or hematologic malignancy | 18 months
  assess the feasibility to enroll patients with a cancer diagnosis or hematologic malignancy
Consent of patients with a cancer diagnosis or hematologic malignancy | 18 months
  assess the feasibility to consent patients with a cancer diagnosis or hematologic malignancy
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by severity | 8 months
  assess the tolerability of psilocybin in patients with a cancer diagnosis or
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by relationship to study treatment. | 8 months
  assess the tolerability of psilocybin in patients with a cancer diagnosis or
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by duration. | 8 months
  assess the tolerability of psilocybin in patients with a cancer diagnosis or
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by seriousness. | 8 months
  assess the tolerability of psilocybin in patients with a cancer diagnosis or
Number of adverse events (AEs) and serious adverse events (SAEs) characterized by type. | 8 months
  assess the tolerability of psilocybin in patients with a cancer diagnosis or

CONTACTS AND LOCATIONS:
Overall Officials: Anna Beck, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No